CLINICAL TRIAL: NCT03192904
Title: Comparison of Energy Instruments and Stapling Device to Dissect Intersegmental Plane in Segmentectomy: A Randomized Controlled Trial
Brief Title: Comparison of Energy Instruments and Stapling Device to Dissect Intersegmental Plane in Segmentectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: One treatment policy showed an advantage at a very high significance level.
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTS-004
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Segmentectomy
Keywords: Lung cancer; Segmentectomy; Postoperative Complication; Stapling Device; Energy Device
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy Instruments Group (Experimental): All enrolled patients will accept robot-assisted or uniportal segmentectomy. After cutting off the relevant segmental arteries and veins, we clamp the segmental bronchus, and then the diseased lung will be ventilated to identify the border of segment according to the collapse region. We use energy instruments dissect intersegmental plane along the determined border. If fast-frozen pathology confirms lung cancer, we will do lymphadenectomy. At last, a drainage tube will be placed.
  Interventions: Device: Energy Instruments
- Stapling Device Group (Experimental): All enrolled patients will accept robot-assisted or uniportal segmentectomy. After cutting off the relevant segmental arteries and veins, we clamp the segmental bronchus, and then the diseased lung will be ventilated to identify the border of segment according to the collapse region. We use stapling device to dissect intersegmental plane along the determined border. If fast-frozen pathology confirms lung cancer, we will do lymphadenectomy. At last, a drainage tube will be placed.
  Interventions: Device: Stapling Device

INTERVENTIONS:
Device: Energy Instruments — Energy Instruments, including electrocautery, harmonic scalpel and LigaSure.
  Arms: Energy Instruments Group
Device: Stapling Device — Stapling Device, including linear stapler and curved stapler.
  Arms: Stapling Device Group

SUMMARY:
According to published studies, there are two main approaches in the dissection of intersegmental plane: stapling devices and energy instrument separation. However, only a few retrospective studies focused on the perioperative outcomes of these two approaches, and there has been no definitive conclusion about which method is better. So the investigators want to conduct a prospective study, trying to figure out this problem.

DETAILED DESCRIPTION:
Lung cancer has been one of the most serious life-threatening diseases of human society. It has the highest morbidity and mortality worldwide among all the malignant tumors. Due to the popularization of low-dose CT and other means of examination, more and more patients with lung cancer are detected in the early phase of disease. Anatomical segmentectomy is one of the standard surgical procedures for these small pulmonary nodules or ground glass opacity (GGO), which are clinically highly suspected or puncture confirmed early lung cancer lesions. Dissection of the intersegmental plane in segmentectomy is a difficulty that have puzzled thoracic surgeons for decades because of the complicated anatomic relationship and variations, along with lack of boundary between pulmonary segments. There are two main approaches in the dissection of intersegmental plane: stapling devices and energy instrument separation. However, only a few retrospective studies focused on the perioperative outcomes of these two approaches in segmentectomy, not to mention in robot assisted segmentectomy, and there has been no definitive conclusion about which method is better. So the investigators want to conduct a prospective study, trying to figure out this problem.

The investigators set incidence rate of postoperative complications as their primary endpoint. According to their calculation, a total of 136 patients will be enrolled (each group has 68 patients).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 70 years old; 2. Pulmonary nodules or GGO found in chest CT examination, and conform with indications for segmentectomy mentioned in NCCN guidelines:

  1. Poor pulmonary reserve or other major comorbidity that contraindicates lobectomy;
  2. Peripheral nodule ≤2 cm with at least one of the following:

  <!-- -->

  1. Pure (Adenocarcinoma in situ) AIS histology;
  2. Nodule has ≥50% ground-glass appearance on CT;
  3. Radiologic surveillance confirms a long doubling time (≥400 days). 3. Normal in preoperative tests, such as blood routine examination, liver function, renal function, coagulation function, etc.

  4. ASA score: Grade I-III. 5. Patients who can coordinate the treatment and research and sign the informed consent.

Exclusion Criteria:

* 1. Patients have history of malignant tumor, or have accepted neoadjuvant chemotherapy and(or) radiotherapy.

  2. Patients have comorbidities in cardiovascular, kidney, lung or hematopoietic system, who cannot tolerate the surgery.

  3. Psychiatric patients。 4. Patient have history of chest trauma or surgery on ipsilateral chest.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD, PhD, Principal Investigator — Ruijin Hospital; Xingshi Chen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Energy Instruments Group | Stapling Device Group
Started | 35 | 35
Completed | 32 | 33
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Energy Instruments Group | Stapling Device Group | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.4) | 53.3 (10.7) | 52.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 33 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 32 | 33 | 65
Smoking History [Count of Participants; unit: Participants] | 6 | 3 | 9
Comorbidity [Count of Participants; unit: Participants] | 10 | 11 | 21
ASA Grade [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) grade is the most commonly used grading system that predicts morbidity and mortality.
  I: Healthy individual with no systemic disease, MORTALITY 0.05% II: Mild systemic disease not limiting activity, MORTALITY 0.4% III: Severe systemic disease that limits activity but is not incapacitating , MORTALITY 4.5% IV: Incapacitating systemic disease which is constantly life-threatening , MORTALITY 25% V: Moribund, not expected to survive 24 hours with or without surgery , MORTALITY 50%
  Participants
    I | 0 | 3 | 3
    II | 31 | 29 | 60
    III | 1 | 1 | 2
Segments resected [Count of Participants; unit: Participants]
  RS1 | 9 | 5 | 14
  RS2 | 0 | 3 | 3
  RS3 | 2 | 1 | 3
  RS6 | 2 | 4 | 6
  RS8 | 1 | 0 | 1
  RS1+RS2 | 0 | 1 | 1
  RS9+RS10 | 1 | 0 | 1
  RS1a+RS2 | 0 | 2 | 2
  RS1b+RS3 | 0 | 1 | 1
  RS1b+RS3b | 0 | 1 | 1
  RS2b+RS3a | 0 | 1 | 1
  RS8b+RS9 | 1 | 0 | 1
  LS1+2 | 7 | 1 | 8
  LS3 | 1 | 1 | 2
  LS6 | 3 | 1 | 4
  LS9 | 1 | 0 | 1
  LS10 | 0 | 1 | 1
  LS1+2+LS3 | 2 | 4 | 6
  LS4+LS5 | 1 | 3 | 4
  LS6+LS8 | 0 | 1 | 1
  LS7+LS8+LS9+LS10 | 0 | 1 | 1
  LS3c | 1 | 0 | 1
  LS1+2+LS3c | 0 | 1 | 1
Approaches(Video-Assisted Thoracic Surgery or Robotic) [Count of Participants; unit: Participants]
  Video-Assisted Thoracic Surgery | 5 | 10 | 15
  Robotic | 27 | 23 | 50
Height [Mean (Standard Deviation); unit: cm] | 162.9 (6.7) | 164.5 (7.7) | 163.7 (7.2)
Weight [Mean (Standard Deviation); unit: kg] | 60.0 (8.1) | 63.4 (8.7) | 61.7 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Complications
Description: The primary outcome was the incidence of postoperative complications, including air leakage (defined as a rate of air flow >50 mL/min lasting more than 3 days), atelectasis (visible on chest X-rays with complaints), hemorrhage (bloody drainage more than 200 mL for 3 consecutive hours), pulmonary infection (visible on chest X-rays with complaint), and pulmonary embolism (confirmed by CT scan).
Time Frame: postoperative in-hospital stay up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
Participants | 11 | 2
Statistical Analysis 1: Comparison: Energy Instruments Group vs Stapling Device Group; Test type: Superiority; p = 0.004, Chi-squared

2. Secondary Outcome: Incidence Rates of Each Postoperative Complications
Time Frame: postoperative in-hospital stay up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
Participants
  Air leakage | 7 | 1
  Pneumothorax | 3 | 0
  Septic shock | 0 | 1
  Cardiac arrest | 1 | 0
  No complications | 21 | 31

3. Secondary Outcome: Preoperative Lung Function
Time Frame: Baseline.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
L | 2.73 (0.50) | 2.80 (0.74)

4. Secondary Outcome: Postoperative Lung Function at the 3rd Month After Surgery
Time Frame: at the 3rd month after surgery
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
L | 2.25 (0.52) | 2.37 (0.62)

5. Secondary Outcome: Postoperative Hospital Stay
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
days | 4.75 (2.38) | 4.24 (2.00)

6. Secondary Outcome: Postoperative ICU Stay
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
Participants
  With ICU stays | 0 | 1
  Without ICU stays | 32 | 32

7. Secondary Outcome: Duration of Drainage
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
days | 3.91 (2.47) | 3.27 (1.53)

8. Secondary Outcome: Mortality in 30 Days After Surgery
Time Frame: postoperative in-hospital stay up to 30 days
Measure: Number; unit: case
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
case | 0 | 0

9. Secondary Outcome: Drainage Volume of the First Day After Surgery
Description: The duration of chest drainage was different, so we analyzed the drainage volume the first day after surgery of each patient.
Time Frame: First day after surgery
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
Milliliter | 176 (122.53) | 142 (94.98)

10. Secondary Outcome: Daily Air Leakage Volume
Time Frame: During drainage time, up to 4 weeks
Population: Data were not collected. Because we found digital drainage system only collect the air leakage rate but not the air leakage volume
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Duration of Surgery
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
min | 138.4 (35.9) | 143.0 (35.7)

12. Secondary Outcome: Blood Loss During Surgery
Time Frame: During surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
ml | 100 [100 to 100] | 100 [75 to 200]

13. Secondary Outcome: Number of Conversions
Description: Proportion of converting to thoracotomy。
Time Frame: During surgery
Measure: Number; unit: case
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
case | 0 | 0

14. Secondary Outcome: Participants With Malignant Tumors
Time Frame: 2 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
Participants | 27 | 30

15. Secondary Outcome: Medical Costs
Time Frame: During hospital stay, up to 24 weeks
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Energy Instruments Group | Stapling Device Group
Number analyzed (Participants) | 32 | 33
USD
  Cost of medical materials | 4214.6 (1185.4) | 3260.1 (352.6)
  Total medical cost | 11136.2 (1902.0) | 111602.5 (2788.9)

ADVERSE EVENTS:
Time Frame: Three months after surgery.
Description: The adverse events occurred were described.
Arm/Group | Energy Instruments Group | Stapling Device Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Energy Instruments Group (N=32) | Stapling Device Group (N=33)
Septic shock (Infections and infestations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
First, we only used electrocautery to divide intersegmental planes in the energy instrument group. Second, the single-center design might lead to selection bias. Third, oncological outcomes were not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03192904/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03192904/ICF_001.pdf